CLINICAL TRIAL: NCT01932918
Title: The Interaction of Nociceptive Stimulation and Various Antinociceptive Modalities on Ischemia Reperfusion Injury
Brief Title: Antinociceptive Modalities on Ischemia Reperfusion Injury
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201001020R
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: End Stage Liver Disease; Lung Cancer
Keywords: reactive oxygen species; ischemia reperfusion injury
MeSH Terms: conditions — End Stage Liver Disease; Lung Neoplasms; Reperfusion Injury | interventions — Analgesia, Patient-Controlled; Morphine; Ketorolac; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PCA with morphine in liver transplant: Intravenous patient controlled analgesia with morphine was used for postoperative pain control in liver transplant recipients.
  Interventions: Drug: Patient controlled analgesia
- PCA with ketorolac in liver transplant: Patient controlled analgesia with morphine and ketorolac was used for postoperative pain control in liver transplant and thoracic surgery patients.
  Interventions: Drug: Patient controlled analgesia
- Intravenous PCA in thoracic surgery: Intravenous patient controlled analgesia was used for postoperative pain control in thoracic surgery patients.
  Interventions: Drug: Patient controlled analgesia
- PCEA in thoracic surgery: Patient controlled epidural analgesia was used for postoperative pain control in thoracic surgery patients.
  Interventions: Drug: Patient controlled analgesia

INTERVENTIONS:
Drug: Patient controlled analgesia — 1. PCA with morphine in liver transplant:
     Intravenous patient controlled analgesia with morphine was used for postoperative pain control in liver transplant recipients.
  2. PCA with morphine and ketorolac:
     Patient controlled analgesia with morphine and ketorolac was used for postoperative pain control in liver transplant and thoracic surgery patients.
  3. Intravenous PCA in thoracic surgery Intravenous patient controlled analgesia was used for postoperative pain control in thoracic surgery patients.
  4. PCEA in thoracic surgery Patient controlled epidural analgesia was used for postoperative pain control in thoracic surgery patients.
  Other Names: morphine; ketorolac; marcaine

SUMMARY:
Postoperative pain caused by surgery-associated tissue injury is a major concern for all the clinical practitioners. Because it affects multiple systems and induces physiological, immunological and psychological changes. Previous literature showed surgical injury induces a systemic inflammatory metabolic-endocrine response that is proportional to the severity of the surgical stress. In surgeries such as liver transplantation, the patients suffer not only from postoperative pain but also an additional oxidative stress caused by ischemia reperfusion. Previous report have proved that an adequate postoperative pain control improves the recovery and reduces the inflammatory cascade by suppression of physiological and psychological stresses. However, the effect of postoperative pain management on ischemia reperfusion injury is unclear so far. In this three year study, we plan to continue our previous study to test the following two hypothesis: (1) postoperative pain exacerbate remote organ injury caused by ischemia reperfusion, (2) the interaction of different antinociceptive modalities on ischemia reperfusion injury.

DETAILED DESCRIPTION:
Our team focused on the study of reperfusion injury in liver transplantation, lung resection and open heart surgeries which need cardiopulmonary bypass. Previous clinical observation showed the increase of lung water in liver transplant recipients. Some patients may even develop pulmonary edema which not only lengthen intensive care unit stay and hospital stay, but also increase morbidity and mortality. In the hepatic ischemia reperfusion animal model, we proved that the release of large amount of reactive oxygen species play an important part in remote lung injury. If propofol, which possesses free radical scavenger property, is given adequately, the production of reactive oxygen species will decrease thus reducing the extent of remote lung injury. In another clinical study, we found that resuming two lung ventilation from one lung ventilation induces a massive superoxide production, which also could be reduced when using propofol for the maintenance of anesthesia.

Postoperative pain caused by surgery-associated tissue injury is a major concern for all the clinical practitioners. Because it affects multiple systems and induces physiological, immunological and psychological changes. Previous literature showed surgical injury induces a systemic inflammatory metabolic-endocrine response that is proportional to the severity of the surgical stress. In surgeries such as liver transplantation, the patients suffer not only from postoperative pain but also an additional oxidative stress caused by ischemia reperfusion. Previous report have proved that an adequate postoperative pain control improves the recovery and reduces the inflammatory cascade by suppression of physiological and psychological stresses. However, the effect of postoperative pain management on ischemia reperfusion injury is unclear so far. In this three year study, we plan to continue our previous study to test the following two hypothesis: (1) postoperative pain exacerbate remote organ injury caused by ischemia reperfusion, (2) the interaction of different antinociceptive modalities on ischemia reperfusion injury.

In the first part, we plan to use the animal model that we have already established to test if analgesics reduce inflammatory responses and remote lung injury caused by hepatic ischemia and to study if different antinociceptive modalities result in different consequences. In the second part, we will recruit patients receiving liver transplantation, lung resection and open heart surgeries needing cardiopulmonary bypass to study the interaction of nociception and various antinociceptive modalities on ischemia reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease patients scheduled for liver transplantation in National Taiwan University Hospital
* Lung cancer patients scheduled for thoracic surgery in National Taiwan University Hospital

Exclusion Criteria:

* preoperative pulmonary dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage liver disease Lung cancer
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
lung injury score | four days

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Cheng Chan, M.D., Principal Investigator — Department of Anesthesiology, NTUH, Taipei, Taiwan
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Lin TF, Yeh YC, Lin FS, Wang YP, Lin CJ, Sun WZ, Fan SZ. Effect of combining dexmedetomidine and morphine for intravenous patient-controlled analgesia. Br J Anaesth. 2009 Jan;102(1):117-22. doi: 10.1093/bja/aen320. Epub 2008 Nov 5. PMID 18987053